CLINICAL TRIAL: NCT02440815
Title: Multimodal MRI Characteristics of Psychotherapy Response in Late Life Depression
Acronym: PRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROI MH101472
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Major Depressive Disorder
Keywords: Psychotherapy; Problem Solving Therapy (PST); Depression; Major Depression; Major Depressive Disorder; Late Life Depression; Multimodal imaging; Magnetic Resonance Imaging (MRI); Cerebral blood flow; Cortical atrophy; White matter lesion
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Problem Solving Therapy (Other): Problem Solving Therapy (PST) is a brief evidence based psychotherapy that is commonly utilized for treatment of LLD. The problem solving therapy includes 12 weekly in person 50 minute sessions.
  Interventions: Behavioral: Problem Solving Therapy

INTERVENTIONS:
Behavioral: Problem Solving Therapy — Problem Solving Therapy (PST) is a brief evidence based psychotherapy that is commonly utilized for treatment of LLD. The problem solving therapy includes 12 weekly in person 50 minute sessions.

SUMMARY:
The specific focus of this study is to gather data regarding the effects of a psychological therapy known as Problem Solving Therapy (PST) on cerebral blood flow (CBF), cortical gray matter (GM) atrophy, subcortical white matter (WM) lesion burden, and measures of cognitive function in subjects with Late Life Major Depressive Disorder (LLD). This research goal will be achieved by recruiting 110 individuals over the age of 65 with LLD. The primary outcomes will be change in CBF, change in GM atrophy, change in WM lesion, change in cognitive function, and change in depression severity from baseline to the end of 12 weeks of PST.

DETAILED DESCRIPTION:
Study procedures include: 1) Telephone screen, 2) Diagnostic evaluation to determine diagnosis of MDD, 3) Baseline evaluation consisting of medical history, cognitive assessment, and MRIs, 4) Participation in 12 weeks of psychotherapy treatment with assessments of depression severity, and 5) Follow up evaluation at 12 weeks consisting of depression, cognitive function, and post treatment MRIs.

Telephone Screen: Older adults who respond to our recruitment efforts for LLD will be screened by telephone using the Patient Health Questionnaire (PHQ-9) and those who obtain a score of 5 or greater will be scheduled for an eligibility appointment within a week of screening. Anyone who endorses the suicide question (item 9) of the PHQ-9 will be scheduled for a same day appointment, and will be seen by the study investigators. Similarly, other exclusion criteria will be assessed using a structured questionnaire. If participants are interested in other treatment referrals these will be provided.

Diagnostic Evaluation: In this assessment, the investigators consent participants and administer measures that address eligibility [i.e., Structured Clinical Interview for Diagnosis of DSM-IV Disorders (SCID)], the 24 item HDRS, Mini Mental Status Exam (MMSE), Clinical Dementia Rating Scale (CDR). To qualify, LLD participants must obtain a diagnosis of MDD (SCID), have an HDRS score of 20 or higher, a MMSE score of 25 or better, and a CDR of 0.5 or less.. Those who do not qualify for the study and/or who are interested in alternate LLD treatments will be offered referrals for services at the outpatient clinics at UCSF or community resources.

Baseline Assessment: After completion of the diagnostic evaluation and being deemed study eligible, LLD participants will be scheduled for a baseline assessment. At the baseline assessment meeting, the HDRS is administered again to confirm depression severity. The baseline assessment consists of 1) demographics and patient characteristics, 2) neuropsychological testing, and 3) depression and functional outcome measures, and 4) multimodal MRI evaluation.

Participant Characteristics: Demographic data, such as age, gender, race, living conditions, marital status, occupation, and education will be obtained as well as previous psychiatric treatment received. Medical comorbidity will be assessed using the Charlson Comorbidity Index (CCI). Medication use will be assessed using the Alzheimer's Disease Neuroimaging Initiative (ADNI) medication history form. Suicidal ideation will be assessed utilizing the Scale for Suicidal Ideation (SSI). The investigators will utilize a clinician rated measures of lifetime history of depressive episodes and depression treatments, the Duke Social Support Index, and the Functional Activities Questionnaire (FAQ) for exploratory analyses.

Cognitive Functioning: Primary cognitive outcome variables will include: the Digit Symbol Substitution Test, the Boston Naming test, and the Rey Auditory Verbal Learning Test as a measure of memory.

Psychotherapeutic Treatment: Problem Solving Therapy (PST) is a brief evidence based psychotherapy that is commonly utilized for treatment of LLD. The problem solving therapy includes 12 weekly in person 50 minute sessions.

Follow up assessments: At 12 weeks, LLD participants will participate in a follow up evaluation that is identical the baseline assessment of depression, cognitive function, and MRI. The investigators will use total HDRS score to determine response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Current DSM-IV diagnosis of MDD, unipolar type, without psychotic features and 6 weeks minimum duration of current depressive episode.
2. Moderate severity of depression using the Hamilton Depression Rating Scale (HDRS > 20).
3. English speaking, male or female
4. 65 years of age or older
5. Good general health
6. Able to give informed consent

Exclusion Criteria:

1. Antidepressant use or psychotherapy within the past 6 weeks or electroconvulsive therapy within the past 6 months.
2. Recent history (<6 months) of substance or alcohol abuse or dependence (DSM-IV criteria).
3. Use of cognitive enhancing medications.
4. Current diagnosis of Post-Traumatic Stress Disorder or other Axis 1 psychiatric disorder.
5. Neurological diseases (e.g., Parkinson's disease, epilepsy, cortical stroke, Alzheimer's disease, traumatic brain injury) or dementia.
6. History of surgical procedures affecting study outcomes.
7. Contraindications for MR exam, i.e., no claustrophobia, no paramagnetic metal implants, able to fit in the MRI machine comfortably (BMI ≤ 38).
8. Acute or uncontrolled medical illness or medication use impacting cognitive function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Rate of change in Cerebral Blood Flow (CBF) as measured by cortical surface-based analysis | Baseline, after 12 weeks of psychotherapy
  CBF will be measured using multimodal MRI processing (individual 2D pseudo ASL image frames). We will pursue a cortical surface-based analysis approach which allows for better spatial normalization of cortical data compared to voxel-based approaches.
Rate of change in Cortical Gray Matter (GM) Atrophy as measured by the FreeSurfer image analysis suite | Baseline, after 12 weeks of psychotherapy
  Cortical Gray Matter Atrophy will be measured using multimodal MRI processing (T1-MRI FreeSurfer image analysis suite version 5.1).
Rate of change in Subcortical White Matter Lesion as measured by WML-T2 FLAIR | Baseline, after 12 weeks of psychotherapy
  Subcortical White Matter Lesion will be measured using multimodal MRI processing [structural T2-weighted Fluid Attenuated Inversion Recovery (FLAIR)].
Rate of change in Depression Severity as measured by the Hamilton Depression Rating Scale (24 item). | Baseline, after 12 weeks of psychotherapy
Rate of change in neuropsychological measures of executive function as measured by the Digit Symbol Substitution Test using total correct | Baseline, after 12 weeks of psychotherapy
Rate of change in expressive language as measured by the Boston Naming Test using total correct. | Baseline, after 12 weeks of psychotherapy
Rate of change in learning and memory as measured by the Rey Auditory Verbal Learning Test using total correct and delayed recall. | Baseline, after 12 weeks of psychotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Scott Mackin, PhD, Principal Investigator — UCSF Department of Psychiatry
Locations (1):
- University of California, San Francisco, Langley Porter Psychiatric Institute, San Francisco, California, United States